CLINICAL TRIAL: NCT02674295
Title: An Open-label, Single-dose Mass Balance Study With a Microtracer Dose of 14C-esketamine in Healthy Male Subjects
Brief Title: A Mass Balance Study With a Microtracer Dose of 14C-esketamine in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108107; 54135419TRD1016 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-02-03; First posted 2016-02-04 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; JNJ-54135419; Esketamine
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): 50 milligram (mg) of oral esketamine, fortified with a microtracer dose of 14C-esketamine, as an aqueous solution mixed with apple juice for administration.
  Interventions: Drug: Esketamine 50 mg
- Cohort 2 (Experimental): 20 mg of intravenous esketamine in 30 milliliter (mL), fortified with a microtracer dose of 14C-esketamine, as a 30-minute intravenous infusion.
  Interventions: Drug: Esketamine 20 mg

INTERVENTIONS:
Drug: Esketamine 50 mg — 50 mg of oral esketamine, fortified with a microtracer dose of 14C-esketamine, as an aqueous solution mixed with apple juice for administration (80 mL total volume)
  Arms: Cohort 1
Drug: Esketamine 20 mg — 20 mg of intravenous esketamine in 30 mL, fortified with a microtracer dose of 14C-esketamine, as a 30-minute intravenous infusion.
  Arms: Cohort 2

SUMMARY:
The purpose of this study is to determine the metabolic disposition of radiolabeled esketamine administered by the oral and intravenous routes in healthy male participants.

DETAILED DESCRIPTION:
This is a single-center, open-label (identity of study drug will be known to participant and study staff), single-dose, parallel-group study. The study consist of Screening Phase (Days -21 to -2), Open-label treatment Phase (Day -1 up to Day 8) and End of Study (9 to 13 days after last study assessment). The total duration of study from the Screening Phase through Follow-up, is 37-41 days. Participants will be assigned to 1 of the two groups (Cohort 1 and Cohort 2) during the treatment phase. The participants will be primarily evaluated to determine the metabolic disposition of radiolabeled esketamine administered by the oral and intravenous routes. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to adhere to the prohibitions and restrictions specified in the protocol
* If a man who is sexually active with a woman of child-bearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the investigator (example, vasectomy, double-barrier, partner using effective contraception) for 3 months following administration of study drug
* Participants with body mass index (BMI) between 18 and 30 kilogram per square meter (kg/m^2) (inclusive), and body weight not less than 50 kg
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic. Note: Average from 3 supine measurements will be used at screening visit
* A 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function, including: Sinus rhythm; Heart rate between 45 and 90 beats per minute (bpm); QTc interval less than or equal to (<=)450 milliseconds (ms); QRS interval of <110 ms; PR interval <200 ms; Morphology consistent with healthy cardiac conduction and function

Exclusion Criteria:

* Participants diagnosed with a current or previous psychiatric or bipolar disorder, as assessed by the investigator, will not be permitted to participate in the study
* Current suicidal or homicidal ideation/intent/behavior as assessed by Columbia Suicide Severity Rating Scale (C-SSRS) at screening
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or at admission to the study center on Day -1 as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs or 12-lead ECG at screening or Day -1, and as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements) within 14 days before study drug administration is scheduled, except for acetaminophen

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Characterisation and Identification of 14C-esketamine Metabolites (Metabolic Profile) | upto 168 hour post-dose
  Collection of urine and feces for 7 days is considered appropriate to characterize the metabolic profile of esketamine. Accelerator mass spectrometry (AMS), an ultrasensitive technique particularly suited for detection of low levels of 14C, will be used to assess levels of the microtracer in whole blood, plasma, and excreta (urine, feces). Plasma, urine and feces selected samples with relatively high radioactive content will be analyzed for metabolic profiling and identification using ultra performance liquid chromatography (UPLC) and AMS.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) or Serious Adverse Events | up to 41 days
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Madison, Wisconsin, United States